CLINICAL TRIAL: NCT04612257
Title: A Pilot Study to Assess Closed-loop Insulin Delivery to Regulate Glucose Levels in Children With Type 1 Diabetes in Outpatient Free-living Settings.
Brief Title: Assessing Closed-loop Insulin Delivery in Children With Type 1 Diabetes.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The sponsor has requested to end the study prematurely due to the accumulation of delays caused by COVID-19 as potential participants were hesitant to allow staff members into their homes or stay at the hospital per the study design.
Sponsor: McGill University (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-5584
Record Dates: First submitted 2020-10-27; First posted 2020-11-02 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Pediatric; Artificial Pancreas
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: The pilot study aims to enroll 20 children participants with type 1 diabetes mellitus using insulin pump therapy. Each participant will undergo a 40-hour intervention period, with the possibility of being invited to a second 40-hour intervention period using the same system.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Insulin alone closed-loop (Experimental): Insulin alone closed-loop algorithm in children with type 1 diabetes in a free-living study.
  Interventions: Other: Insulin-alone closed-loop

INTERVENTIONS:
Other: Insulin-alone closed-loop — 40-hour intervention period using the insulin-alone closed-loop system.

SUMMARY:
The objective of this clinical trial is to assess the safety of our insulin dosing algorithm in children with type 1 diabetes in a free-living study.

DETAILED DESCRIPTION:
This is a preliminary pilot study to generate data to optimize an insulin dosing algorithm to regulate glucose levels in children with type 1 diabetes. There will be up to two 40-hour test in outpatient settings, in which we will assess an insulin dosing algorithm. The two tests will allow us to compare different tunings in the same patient (this allows easier interpretation of the data). For example, if in a specific participant, the dosing algorithm reduced insulin delivery at night to avoid low blood glucose levesl but led to a rebound increase in glucose levels, then a second visit with a slightly different target range will help answer this question. The objective of this clinical trial is to assess the safety of our algorithm in children with type 1 diabetes in a free-living study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female children between 2 and 13 years of age.
2. Clinical diagnosis of type 1 diabetes mellitus (the diagnosis of type 1 diabetes is based on the investigator's judgment).
3. Using insulin pump therapy for at least 3 months
4. For participants aged 7-13 years: Total daily insulin dose ≤ 40 units and 0.5 ≥ units/kg/day. For participants aged 2-6 years: Total daily insulin dose [8, 40] units and 0.3 ≥ units/kg/day.
5. Most recent (in the last 6 months) HbA1c ≤ 12%.

Exclusion Criteria:

1. Using Medtronic 670G automated insulin delivery system (since participant's basal rates and insulin-to-carbohydrate ratios may reflect the use of 670G; generally overestimated by 20%).
2. Severe hypoglycaemia or ketoacidosis episode ≤ two months before admission.
3. Medical illness or other issues likely to interfere with study participation or with the ability to complete the trial by the judgment of the investigator.

Ages: 2 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-06-13 (Actual)

PRIMARY OUTCOMES:
Time in range | 40-hour intervention
  Percentage of time of glucose levels spent in the target range (3.9-10.0 mmol/L).

SECONDARY OUTCOMES:
Specific time in range | 40-hour intervention
  Percentage of time of glucose levels spent a. between 3.9 and 7.8 mmol/L; b. below 3.9 mmol/L; c. below 3.3 mmol/L; d. below 2.8 mmol/L; e. above 10.0 mmol/L; f. above 13.9 mmol/L; g. above 16.7 mmol/L.
Specific nighttime time in range | 40-hour intervention
  Percentage of time (00:00-6:00) of glucose levels spent a. below 3.9 mmol/L; b. between 3.9 and 7.8 mmol/L; c. between 3.9 and 10.0 mmol/L; d. below 3.3 mmol/L; e. below 2.8 mmol/L; f. above 10.0 mmol/L; g. above 13.9 mmol/L; h. above 16.7 mmol/L.
Mean glucose levels | 40-hour intervention
  Mean glucose levels.
Standard deviation of glucose levels and insulin delivery | 40-hour intervention
  Standard deviation of glucose levels and insulin delivery.
Coefficient of variance of glucose levels and insulin delivery | 40-hour intervention
  Coefficient of variance of glucose levels and insulin delivery.
Total insulin delivery | 40-hour intervention
  Total amount of insulin delivered.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Legault, MD, Principal Investigator — Montreal Children's Hospital of the MUHC
Locations (1):
- McGill University Health Centre Research Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pickup JC, Keen H, Parsons JA, Alberti KG. Continuous subcutaneous insulin infusion: an approach to achieving normoglycaemia. Br Med J. 1978 Jan 28;1(6107):204-7. doi: 10.1136/bmj.1.6107.204. PMID 340000
- [Background] Thabit H, Tauschmann M, Allen JM, Leelarathna L, Hartnell S, Wilinska ME, Acerini CL, Dellweg S, Benesch C, Heinemann L, Mader JK, Holzer M, Kojzar H, Exall J, Yong J, Pichierri J, Barnard KD, Kollman C, Cheng P, Hindmarsh PC, Campbell FM, Arnolds S, Pieber TR, Evans ML, Dunger DB, Hovorka R. Home Use of an Artificial Beta Cell in Type 1 Diabetes. N Engl J Med. 2015 Nov 26;373(22):2129-2140. doi: 10.1056/NEJMoa1509351. Epub 2015 Sep 17. PMID 26379095
- [Background] Wasserman DH, Zinman B. Exercise in individuals with IDDM. Diabetes Care. 1994 Aug;17(8):924-37. doi: 10.2337/diacare.17.8.924. No abstract available. PMID 7956645
- [Background] Tauschmann M, Allen JM, Nagl K, Fritsch M, Yong J, Metcalfe E, Schaeffer D, Fichelle M, Schierloh U, Thiele AG, Abt D, Kojzar H, Mader JK, Slegtenhorst S, Barber N, Wilinska ME, Boughton C, Musolino G, Sibayan J, Cohen N, Kollman C, Hofer SE, Frohlich-Reiterer E, Kapellen TM, Acerini CL, de Beaufort C, Campbell F, Rami-Merhar B, Hovorka R; KidsAP Consortium. Home Use of Day-and-Night Hybrid Closed-Loop Insulin Delivery in Very Young Children: A Multicenter, 3-Week, Randomized Trial. Diabetes Care. 2019 Apr;42(4):594-600. doi: 10.2337/dc18-1881. Epub 2019 Jan 28. PMID 30692242
- [Background] Del Favero S, Boscari F, Messori M, Rabbone I, Bonfanti R, Sabbion A, Iafusco D, Schiaffini R, Visentin R, Calore R, Moncada YL, Galasso S, Galderisi A, Vallone V, Di Palma F, Losiouk E, Lanzola G, Tinti D, Rigamonti A, Marigliano M, Zanfardino A, Rapini N, Avogaro A, Chernavvsky D, Magni L, Cobelli C, Bruttomesso D. Randomized Summer Camp Crossover Trial in 5- to 9-Year-Old Children: Outpatient Wearable Artificial Pancreas Is Feasible and Safe. Diabetes Care. 2016 Jul;39(7):1180-5. doi: 10.2337/dc15-2815. Epub 2016 May 10. PMID 27208335
- [Background] DeBoer MD, Breton MD, Wakeman C, Schertz EM, Emory EG, Robic JL, Kollar LL, Kovatchev BP, Chernavvsky DR. Performance of an Artificial Pancreas System for Young Children with Type 1 Diabetes. Diabetes Technol Ther. 2017 May;19(5):293-298. doi: 10.1089/dia.2016.0424. Epub 2017 Apr 20. PMID 28426239
- [Background] Gingras V, Rabasa-Lhoret R, Messier V, Ladouceur M, Legault L, Haidar A. Efficacy of dual-hormone artificial pancreas to alleviate the carbohydrate-counting burden of type 1 diabetes: A randomized crossover trial. Diabetes Metab. 2016 Feb;42(1):47-54. doi: 10.1016/j.diabet.2015.05.001. Epub 2015 Jun 10. PMID 26072052
- [Background] Taleb N, Emami A, Suppere C, Messier V, Legault L, Ladouceur M, Chiasson JL, Haidar A, Rabasa-Lhoret R. Efficacy of single-hormone and dual-hormone artificial pancreas during continuous and interval exercise in adult patients with type 1 diabetes: randomised controlled crossover trial. Diabetologia. 2016 Dec;59(12):2561-2571. doi: 10.1007/s00125-016-4107-0. Epub 2016 Oct 4. PMID 27704167
- [Background] Haidar A, Messier V, Legault L, Ladouceur M, Rabasa-Lhoret R. Outpatient 60-hour day-and-night glucose control with dual-hormone artificial pancreas, single-hormone artificial pancreas, or sensor-augmented pump therapy in adults with type 1 diabetes: An open-label, randomised, crossover, controlled trial. Diabetes Obes Metab. 2017 May;19(5):713-720. doi: 10.1111/dom.12880. Epub 2017 Mar 8. PMID 28094472
- [Background] Gingras V, Haidar A, Messier V, Legault L, Ladouceur M, Rabasa-Lhoret R. A Simplified Semiquantitative Meal Bolus Strategy Combined with Single- and Dual-Hormone Closed-Loop Delivery in Patients with Type 1 Diabetes: A Pilot Study. Diabetes Technol Ther. 2016 Aug;18(8):464-71. doi: 10.1089/dia.2016.0043. Epub 2016 May 18. PMID 27191385
- [Result] Haidar A, Legault L, Matteau-Pelletier L, Messier V, Dallaire M, Ladouceur M, Rabasa-Lhoret R. Outpatient overnight glucose control with dual-hormone artificial pancreas, single-hormone artificial pancreas, or conventional insulin pump therapy in children and adolescents with type 1 diabetes: an open-label, randomised controlled trial. Lancet Diabetes Endocrinol. 2015 Aug;3(8):595-604. doi: 10.1016/S2213-8587(15)00141-2. Epub 2015 Jun 8. PMID 26066705
- [Result] Haidar A, Rabasa-Lhoret R, Legault L, Lovblom LE, Rakheja R, Messier V, D'Aoust E, Falappa CM, Justice T, Orszag A, Tschirhart H, Dallaire M, Ladouceur M, Perkins BA. Single- and Dual-Hormone Artificial Pancreas for Overnight Glucose Control in Type 1 Diabetes. J Clin Endocrinol Metab. 2016 Jan;101(1):214-23. doi: 10.1210/jc.2015-3003. Epub 2015 Nov 2. PMID 26523526